CLINICAL TRIAL: NCT07003685
Title: Efficacy and Safety of Posterior Chamber Glaucoma Drainage Device in Refractory Pseudophakic Glaucoma Patients
Brief Title: Efficacy and Safety of Posterior Chamber Glaucoma Drainage Device
Acronym: AGV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital of Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Quyen Vo Mai Huynh, Vice Head of General Planning Department, Eye Hospital of Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 320/BVM-HDDD
Record Dates: First submitted 2025-06-03; First posted 2025-06-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Anterior chamber (Active Comparator): Control group
  Interventions: Device: GDD in aterior chamber
- Study group (Experimental): AGV in Posterior chamber
  Interventions: Device: GDD in posterior chamber

INTERVENTIONS:
Device: GDD in posterior chamber — GDD in posterior chamber
  Arms: Study group
Device: GDD in aterior chamber — GDD in anterior chamber
  Arms: Anterior chamber

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Ahmed glaucoma valve (AGV) implantation in the posterior chamber (ciliary sulcus) compared with the traditional anterior chamber placement in patients with refractory pseudophakic glaucoma, who are adults (>18 years), have undergone cataract surgery with intraocular lens implantation, and are unresponsive to maximal medical therapy.

The main questions it aims to answer are:

Does posterior chamber AGV implantation effectively lower intraocular pressure (IOP) compared to anterior chamber implantation? Does posterior chamber AGV implantation result in less corneal endothelial cell loss and lower rates of postoperative complications compared to anterior chamber implantation?

Researchers will compare the two groups:

Intervention group: AGV implantation in the posterior chamber (ciliary sulcus) Control group: AGV implantation in the anterior chamber

Participants will:

Undergo a baseline evaluation, including ocular examination, IOP measurement, corneal endothelial cell density (ECD) and variability, visual field testing, and optic nerve imaging.

Be randomized into two groups based on a computer-generated randomization method.

Receive either posterior chamber or anterior chamber AGV implantation. Be followed postoperatively at specified intervals (1 day, 1 week, 1 month, 3 months, 6 months, 12 months) for IOP, use of glaucoma medications, visual acuity (Snellen, logMAR), corneal ECD, and endothelial cell variability (CV).

Undergo regular assessments for postoperative complications such as hypotony, choroidal detachment, hyphema, infection, and device-related issues.

Provide informed consent after explanation of potential risks and benefits of the procedure.

This study will use a prospective, randomized controlled clinical trial design, enrolling at least 29 eyes in each group, conducted at the Glaucoma Department of Ho Chi Minh City Eye Hospital from March 2024 to March 2027

DETAILED DESCRIPTION:
1. Background and Rationale Refractory glaucoma in pseudophakic eyes presents a significant clinical challenge due to its resistance to maximal medical therapy and often poor response to conventional filtering surgeries. In these patients, the implantation of a glaucoma drainage device (GDD), such as the Ahmed glaucoma valve (AGV), has emerged as a viable therapeutic strategy. Traditionally, GDDs are inserted with the tube placed into the anterior chamber (AC). However, anterior chamber placement may be associated with long-term complications, such as corneal endothelial decompensation, synechiae, iris chafing, and chronic inflammation.

   The posterior chamber, specifically the ciliary sulcus, offers an alternative site for tube placement in pseudophakic eyes where the natural lens has already been removed. The sulcus location provides a deeper site for the tube, reducing the risk of contact with the corneal endothelium. Preliminary evidence and retrospective series suggest that sulcus placement can achieve comparable IOP-lowering efficacy while minimizing endothelial cell loss. However, to date, there is a lack of high-quality randomized controlled trials that rigorously compare the safety and efficacy outcomes of anterior vs posterior chamber tube placement in pseudophakic patients.

   This study is designed to address this gap in the literature by evaluating Ahmed glaucoma valve implantation with tube placement in the posterior chamber (ciliary sulcus) compared with standard anterior chamber placement in patients with refractory pseudophakic glaucoma.
2. Objectives Primary Objective To evaluate and compare the intraocular pressure (IOP) reduction at 12 months following AGV implantation in the posterior chamber (ciliary sulcus) versus anterior chamber placement in eyes with refractory pseudophakic glaucoma.

   Secondary Objectives To assess the difference in corneal endothelial cell loss between the two groups.

   To compare the number of glaucoma medications required postoperatively. To evaluate the incidence of postoperative complications in both surgical groups.

   To determine the cumulative surgical success rates (complete and qualified success).
3. Study Design This is a prospective, randomized, controlled, interventional clinical trial conducted at the Glaucoma Department of Ho Chi Minh City Eye Hospital. The study will enroll a total of 58 eyes (29 eyes per group), assigned to either anterior or posterior chamber AGV implantation via computer-generated randomization.

   The study period spans from March 2024 to August 2027, including a 12-month follow-up for each participant.
4. Participants

   Eligible participants are adults aged ≥18 years with:

   A diagnosis of refractory glaucoma Pseudophakia (presence of posterior chamber intraocular lens) IOP ≥ 21 mmHg despite maximal tolerated medical therapy No previous glaucoma drainage device implantation in the study eye Patients with active uveitis, neovascular glaucoma, corneal decompensation, or contraindications to surgery will be excluded.
5. Surgical Technique 5.1 Common Steps (Both Groups) General or local peribulbar anesthesia Fornix-based conjunctival flap in the superotemporal quadrant Priming of the AGV device Fixation of the plate 8-10 mm posterior to the limbus using 8-0 nylon sutures 5.2 Anterior Chamber Group Tube trimmed and beveled for anterior chamber entry Insertion through a scleral tunnel into the anterior chamber at the limbus, between iris and cornea Tube coverage with donor scleral patch graft and conjunctival closure 5.3 Posterior Chamber Group Complete anterior vitrectomy via pars plana approach if required to clear vitreous Tube insertion through the sclera into the ciliary sulcus, posterior to the iris and anterior to the IOL Tube secured and covered with a scleral patch graft, followed by conjunctival closure
6. Follow-Up Protocol

   Participants will be followed at:

   Post-op Day 1 Week 1 Month 1, 3, 6, and 12

   At each visit, the following will be assessed:

   IOP (Goldmann applanation) Best corrected visual acuity (Snellen/logMAR) Number of glaucoma medications Corneal endothelial cell density (specular microscopy) Central corneal thickness Slit-lamp biomicroscopy and funduscopy Recording of adverse events and complications
7. Outcome Measures Primary Outcome Mean IOP at 12 months Secondary Outcomes Change in corneal endothelial cell density Proportion of eyes achieving target IOP (<21 mmHg) without medications (complete success) Proportion achieving target IOP with medications (qualified success) Number of medications required at each follow-up Rates of postoperative complications: hypotony, hyphema, choroidal detachment, corneal decompensation, tube obstruction, infection
8. Data Collection and Management All data will be recorded in standardized case report forms and entered into a secure electronic database. Specular microscopy measurements will be standardized using the same device (Topcon SP-3000P) and operator for all participants. Data quality will be reviewed regularly by the study monitoring committee.
9. Statistical Analysis

   Descriptive statistics will be used to summarize demographics and baseline characteristics. Differences between groups will be assessed using:

   Student's t-test for continuous variables (e.g., IOP, endothelial count) Chi-square or Fisher's exact test for categorical outcomes Kaplan-Meier survival analysis for surgical success P-values <0.05 considered statistically significant
10. Safety Considerations All surgical procedures will be performed by experienced glaucoma surgeons. Standard aseptic and surgical safety protocols will be followed. Any serious adverse event (SAE) will be reported to the Institutional Review Board (IRB) and study monitoring committee.
11. Significance of the Study This study will be the first randomized controlled trial in Vietnam comparing anterior vs posterior chamber Ahmed valve implantation in pseudophakic glaucoma. The results will help guide surgical decision-making in patients at risk of corneal decompensation and improve long-term visual outcomes in this challenging population.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Diagnosis of refractory glaucoma (uncontrolled intraocular pressure despite maximal tolerated antiglaucoma medications).
* History of cataract extraction with intraocular lens implantation (pseudophakia).
* Agreement to participate in the study and ability to comply with outpatient follow-up requirements

Exclusion Criteria:

* Presence of corneal opacities that preclude accurate endothelial assessment.
* Co-existing corneal diseases that could affect endothelial cell status (e.g., Fuchs' dystrophy, corneal edema).
* Single-eye (monocular) status.
* Systemic medical conditions affecting coagulation or carrying increased surgical risk (e.g., uncontrolled diabetes, bleeding disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
IOP | IOP change at 12 months postoperatively
ECD | Corneal endothelial cell density (ECD) change from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Quyen Vo Mai Huynh, M.D., Principal Investigator — Ho Chi Minh city Eye Hospital
Locations (1):
- Hochiminh city Eye Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
IPD are to be shared after the study have been started.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Jun 2025 - Jun 2030
Access Criteria: No criteria